CLINICAL TRIAL: NCT02571387
Title: Study of the Effects of Mindfulness on Impulsive Eating, Motivation Toward Exercise, and Weight Loss in Obese Patients: Randomized Controlled Trial
Brief Title: MindOb: A 12-month Computerized Mindfulness-based Intervention for Obese Individuals
Acronym: MindOb
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Paris 5 - Rene Descartes (Other)
Collaborators: Hospital Ambroise Paré Paris (Other); Nestlé Foundation (Other)
Responsible Party: Principal Investigator, Ruffault Alexis, Doctoral candidate, University of Paris 5 - Rene Descartes
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EA4057-mindob
Record Dates: First submitted 2015-10-02; First posted 2015-10-08 (Estimated); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Obesity; Binge-Eating Disorder
Keywords: Motivation; Impulsive eating; Mindfulness; Self-help; Physical activity; Weight-loss
MeSH Terms: conditions — Obesity; Binge-Eating Disorder; Motor Activity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mindfulness (Experimental): Computerized mindfulness-based intervention. 10 minutes per day, every day for 12 months of MP3 listening. Guidelines are in line with main mindfulness-based interventions (MBSR, MBCT, ACT). Participants can choose between 4 audio recordings (sessions): awareness of the breathing, awareness of postures and bodily sensations, acceptance of thoughts and emotions, and awareness of bodily sensations and related thoughts and emotions while executing 5 squats.
  Interventions: Behavioral: Mindfulness-based intervention
- Sham meditation (Sham Comparator): Computerized sham meditation intervention. 10 minutes per day, every day for 12 months of MP3 listening. The unique guideline is to "meditate" at the beginning of each session. Participants can choose between 4 audio backgrounds: forest, night, beach, and river.
  Interventions: Behavioral: Sham meditation
- Treatment as usual (No Intervention): Usual care in a nutrition pole in France: nutrition, diet, exercise.

INTERVENTIONS:
Behavioral: Mindfulness-based intervention
  Arms: Mindfulness
Behavioral: Sham meditation
  Arms: Sham meditation

SUMMARY:
The purpose of this study is to evaluate the efficacy of a daily 12-month computerized mindfulness-based intervention in obese patients diagnosed with Binge Eating Disorder (BED) on: impulsive eating, motivation toward exercise, and weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged between 18 and 65 years
* Obese (BMI >= 30)
* Recruited from the nutrition pole of Ambroise Paré Hospital
* Diagnosed with Binge-Eating Disorder (BED) according to DSM5 criteria
* Informed consent provided during inclusion interview

Exclusion Criteria:

* Already participating in a clinical trial
* Bariatric surgery patients (except for gastric band removed at least 3 years before)
* Planned bariatric surgery
* Central obese (genetic)
* Pregnant women
* No internet access at home
* Difficulties to understand French language
* Patients under social protection
* Cognitive dysfunctions in understanding simple guidelines provided by the paramedical staff (e.g., diet or exercise guidelines)
* Auditory disorders not allowing to hear audio files
* Blurred vision not allowing to use Internet

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-05; Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Change in impulsive eating (TFEQ-R18 "uncontrolled eating" subscale) | From baseline to study completion (12 months). Assessments at baseline, 1 month, 6 months and 12 months.

SECONDARY OUTCOMES:
Change in motivational regulation toward exercise (BREQ-II) | From baseline to study completion (12 months). Assessments at baseline, 1 month, 6 months and 12 months.
  Behavioral Regulation in Exercise Questionnaire-II (5 subscales): amotivation, external regulation, introjected regulation, identified regulation, intrinsic regulation
Change in self-reported physical activity (IPAQ) | From baseline to study completion (12 months). Assessments at baseline, 1 month, 6 months and 12 months.
  International Physical Activity Questionnaire short form
Change in pedometers-measured physical activity | From baseline to study completion (12 months). Assessments at baseline, 6 months and 12 months.
  Pedometers on a daily basis for 7 days (ref: ONWalk100)
Change in self-reported anxiety and depression (HADS) | From baseline to study completion (12 months). Assessments at baseline, 1 month, 6 months and 12 months.
  Hospital Anxiety and Depression Scale (2 subscales): anxiety and depression
Change in mindfulness skills (MAAS, AAQ-II) | From baseline to study completion (12 months). Assessments at baseline, 1 month, 6 months and 12 months.
  Combination of scores in Mindful Attention Awareness Scale; Acceptance and Action Questionnaire-II
Change in daily mindful responding (DMRS) | From baseline to study completion (12 months). Assessments at baseline, 6 months and 12 months.
  Daily Mindful Responding Scale on a daily basis for 7 days (at baseline, 6 months and 12 months)
Change in plasma concentration of leptin, adiponection and BDNF | From baseline to study completion (12 months). Assessments at baseline, 6 months and 12 months.
Change in body mass index (kg/m2) | From baseline to study completion (12 months). Assessments at baseline, 6 months and 12 months.
  BMI as measured by a physician
Change in food intake | From baseline to study completion (12 months). Assessments at baseline, 6 months and 12 months.
  Dietary survey on a daily basis for 7 days (at baseline, 6 months and 12 months)

OTHER OUTCOMES:
Compliance to the intervention (number of sessions done divided by number of session due) | From baseline to study completion (12 months). Assessments at baseline, 1 month, 6 months and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Czernichow, Pr, Principal Investigator — Hospital Ambroise Paré Paris; Cécile Flahault, PhD, Study Director — University Paris 5 - Rene Descartes
Locations (1):
- Hôpital Ambroise Paré, Assistance Publique-Hôpitaux de Paris, Boulogne-Billancourt, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ruffault A, Carette C, Lurbe I Puerto K, Juge N, Beauchet A, Benoliel JJ, Lacorte JM, Fournier JF, Czernichow S, Flahault C. Randomized controlled trial of a 12-month computerized mindfulness-based intervention for obese patients with binge eating disorder: The MindOb study protocol. Contemp Clin Trials. 2016 Jul;49:126-33. doi: 10.1016/j.cct.2016.06.012. Epub 2016 Jun 29. PMID 27370231
- See also: Academic webpage of the PhD candidate running the study — http://recherche.parisdescartes.fr/LPPS_esl/Membres/Doctorants/Alexis-Ruffault